CLINICAL TRIAL: NCT07370233
Title: Synchronous Percutaneous Facet Radiofrequency and Spinal Fixation With Epidural Injection Therapy as a Management for Persistent Radicular Pain After Microdiscectomy
Brief Title: Triple Therapy Strategy for Managing Persistent Pain After Spinal Microdiscectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Adel Farag Al Kholy, Professor of Medical Biochemistry, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rc 8-1-2023
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Spinal Disk Injury
MeSH Terms: interventions — Injections, Epidural; Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple Therapy Group (Active Comparator): Patients with failed back surgery syndrome who receive a combined intervention consisting of thermal radiofrequency ablation of the medial branch, percutaneous spinal fixation (Sextant system), and an epidural injection of triamcinolone mixed with hyaluronidase.
  Interventions: Drug: Epidural Injection; Procedure: thermal Radiofrequency Ablation; Procedure: Spinal Fixation; Diagnostic Test: ELISA
- Spinal Fixation Only (Active Comparator): Patients with failed back surgery syndrome who undergo percutaneous spinal fixation only, using the Sextant system to stabilize the adjoining vertebrae.
  Interventions: Procedure: Spinal Fixation; Diagnostic Test: ELISA
- Healthy Control (Active Comparator): A cross-matched group of healthy volunteers used solely as a baseline reference for serum inflammatory cytokine levels.
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Drug: Epidural Injection — Advanced Touhy needle delivery of 80 mg triamcinolone and 1500 IU hyaluronidase into the epidural space to target inflammation and adhesions
  Arms: Triple Therapy Group
Procedure: thermal Radiofrequency Ablation — Thermal denervation of the medial branch of the facet nerve at 80°C for 120 seconds using an 18-gauge insulated RF needle.
  Arms: Triple Therapy Group
Procedure: Spinal Fixation — Percutaneous insertion of polyaxial screws and pre-contoured rods via the Sextant System to stabilize the affected spinal levels.
  Arms: Spinal Fixation Only; Triple Therapy Group
Diagnostic Test: ELISA — Collection of blood samples (S1 at booking and S2 at 6 months) for ELISA estimation of serum biomarkers including TNF-α, IL-1β, and IL-6.

SUMMARY:
This interventional study evaluates a "triple therapy" approach-combining percutaneous spinal fixation, facet radiofrequency ablation, and epidural steroid/hyaluronidase injection-for patients with Failed Back Surgery Syndrome (FBSS). The study compares this combined strategy against spinal fixation alone to determine its effectiveness in reducing chronic radicular pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent back pain after microdiscectomy (FBSS).
* Failure of conservative treatment for at least six months.
* Positive results on a diagnostic lumbar facet nerve block.

Exclusion Criteria:

* Spinal instability, fractures, or spondylolisthesis.
* Severe psychiatric disorders.
* Baseline ODI score higher than 60%.
* Opioid users or history of adverse reactions to steroids.

Ages: 23 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (NRS) | 6 months post-intervention
  Assessment of back and radicular pain using the 10-point Numeric Rating Scale (NRS)(Score on a scale of 0 to 10)
Change in Disability Level (ODI) | 6 months post-intervention
  Measurement of functional disability using the Oswestry Disability Index (ODI).

SECONDARY OUTCOMES:
Serum Concentration of Pro-inflammatory Cytokines (TNF-α) | 6 months post-intervention
  Evaluation of the anti-inflammatory mechanism by measuring serum Tumor Necrosis Factor-alpha levels via ELISA.

OTHER OUTCOMES:
Success Rate of Pain and Disability Mitigation | 6 months post-intervention
  : The percentage of participants achieving a successful treatment outcome at 6 months. Success is defined as an "Excellent" or "Good" grade according to Odom's criteria, indicating significant improvement or minimal persistence of preoperative symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shible, MD, Principal Investigator — Lecturer at Department of Orthopedic Surgery, Faculty of Medicine; Adel Samy Elhammady, MD, Principal Investigator — Lecturer at Department of Orthopedic Surgery, Faculty of Medicine
Locations (1):
- Faculty of Medicine, Benha University, Banhā, Qalyubia Governorate, Egypt